CLINICAL TRIAL: NCT06013644
Title: Comparative Efficacy of Acupuncture, Dry Needle and Botox Injection in Management of Patient With Myofascial Pain Dysfunction Syndrome Using Electromyography and Visual Analogue Scale: A Randomized Clinical Trial
Brief Title: Acupuncture, Dry Needle and Botox Injection in Management of Patient With Myofascial Pain Dysfunction Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wajmah Sayed Karim Al Sayed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17223
Record Dates: First submitted 2023-07-07; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Myofascial Trigger Point Pain; Myofascial Pain Syndrome
Keywords: botox injection; dry needle; myofascial trigger point pain; acupuncture
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acupuncture needle (study group A) (Active Comparator): a weekly session for 4-6 weeks on needle for each acupoint for at least 20 minutes the included acupoints are ST6, ST7, SI 18, ST 19, GB 2
  Interventions: Device: Acupuncture needle
- Dry needle (study group B) (Active Comparator): a weekly session for 4-6 weeks the trigger point is held by thumb and index fingers and the needle approaches the point perpendicular to the skin and rotated clockwise for 2-3 minutes
  Interventions: Device: Dry needle
- Botox injection (study group C) (Active Comparator): each patient will receive a one time treatment of a suitable dose (estimated by the research team) according to the severity of the symptoms
  Interventions: Drug: Botox Injectable Product

INTERVENTIONS:
Device: Acupuncture needle — a weekly session for 4-6 weeks on needle for each acupoint for at least 20 minutes the included acupoints are ST6, ST7, SI 18, ST 19, GB 2
  Arms: Acupuncture needle (study group A)
Device: Dry needle — a weekly session for 4-6 weeks the trigger point is held by thumb and index fingers and the needle approaches the point perpendicular to the skin and rotated clockwise for 2-3 minutes
  Arms: Dry needle (study group B)
Drug: Botox Injectable Product — each patient will receive a one time treatment of a suitable dose (estimated by the research team) according to the severity of the symptoms
  Arms: Botox injection (study group C)

SUMMARY:
Evaluating myofascial pain dysfunction symptoms using acupuncture, dry needle and Botox injection using electromyography and visual Analogue Scale on two time intervals at 2 and 6 months after the intervention

DETAILED DESCRIPTION:
All the patients will be selected and examine from the outpatient clinic of Oral and Maxillofacial surgery department. Faculty of Dentistry, Cairo University, Egypt.

Electromyography examination will be conducted in the department of neurophysiology department. faculty of Medicine, Cairo University, Egypt. Adult patients of both sexes, aged from 15 to 60 years with myofascial pain dysfunction syndrome complaining from sign and symptoms of pain or muscles spams and examination shows trigger points in masticatory muscles. selected patients must have not received any other form of surgical treatment related to TMJ disorders All patients involved in this study will be divided into three groups, each group will receive a technique for one side of MPDS, involving acupuncture, dry needle, and Botox injection.

for both, acupuncture group and dry needling group, patients should receive a session/week for 4-6 weeks

ELIGIBILITY:
Accepts Healthy Volunteers

Inclusion Criteria:

* Healthy Volunteers
* MPDS patient
* Adult patients of both sexes, aged from 15 to 60 years
* signs and symptoms of pain or muscles spams
* Trigger points in masticatory muscles
* Patients had not received any other form of surgical treatment related to TMJ disorders
* Cooperative patient

Exclusion Criteria:

* Severe bleeding tendency, e.g. anticoagulant therapy, thrombocytopenia
* Edentulous patients, and total dental prosthesis.
* Psychologically disturbed and mental disturbance patients
* major systemic disorders (- Valvular heart disease: avoid indwelling needles)
* seizure patients
* A confirmed or suspected diagnosis of an inflammatory disorder and autoimmune.
* Patient on Medication (insulin- corticosteroids, nonsteroidal anti-inflammatory therapy or narcotics, muscle relaxants, herbal medicines.)
* Analgesic or anti-depressants over the last 2 weeks.
* Any anatomical abnormality in TMJ.
* Pregnant women.
* Allergies to metals.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
change of electrical activity of mastication muscles from the baseline measurement | 2 months after treatment
  change of electrical activity of mastication muscles from the baseline measurement through assessment of muscle tone using electromyography (EMG) in microvolts and refer to the behavior of muscles: at (rest /open, chewing, clenching)
change of electrical activity of mastication muscles from the baseline measurement | 6 months after treatment
  change of electrical activity of mastication muscles from the baseline measurement through assessment of muscle tone using electromyography (EMG) in microvolts and refer to the behavior of muscles: at (rest /open, chewing, clenching)

SECONDARY OUTCOMES:
change of Pain perception from baseline measurement during maximum mouth opening in millimetres and rest by a Visual Analog Score (where Zero means no pain and 10 means the worst pain possible) | 2 months after treatment
  change of Pain perception from the baseline measurement during maximum mouth opening in millimetres and rest by a Visual Analog Score (where Zero means no pain and 10 means the worst pain possible)
change of Pain perception from baseline measurement during maximum mouth opening in millimetres and rest by a Visual Analog Score (where Zero means no pain and 10 means the worst pain possible) | 6 months after treatment
  change of Pain perception from the baseline measurement during maximum mouth opening in millimetres and rest by a Visual Analog Score (where Zero means no pain and 10 means the worst pain possible)

OTHER OUTCOMES:
Patient Satisfaction questionnaire | 2 months after treatment
  Score of 1 to 10 where (1 means least satisfaction and 10 means most satisfaction
Patient Satisfaction questionnaire | 6 months after treatment
  Score of 1 to 10 where (1 means least satisfaction and 10 means most satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Wajma Sayed Karim Al Sayed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
All the study data will be available upon publication after completion of the study